CLINICAL TRIAL: NCT05361603
Title: Acceptability of Simultaneous Screening for Viral Hepatitis B, C and HIV Among Drug Users in Non-conventional Facilities "Outside the Walls" Using the Dual Screening Method TROD (Rapid Diagnostic Tests) and FibroScan
Brief Title: Acceptability of Simultaneous Screening for Viral Hepatitis B, C and HIV Among Drug Users in Non-conventional Structures
Acronym: SCANVIR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I17011_SCANVIR
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis C; Transmission, Intravenous Drug Abuser; Addiction, Alcohol; Addiction Opiate; Hepatitis C Virus Infection, Response to Therapy of
Keywords: hepatitis C; Elimination; HBV; HIV; PWID; Addiction; Care structure
MeSH Terms: conditions — Hepatitis C; Alcoholism; Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The principle is to propose dedicated monthly screening days bringing together the health personnel involved (hepatologist, addictologist, nurse in charge of the program, addictology nurse and social worker) and to propose appropriate management for each situation assessed.

DETAILED DESCRIPTION:
1. Information on screening, the days are announced by :

   * Mailing to health professionals in the Haute-Vienne Department,
   * Announcement to the different professional orders concerned (doctors, pharmacists, midwives, nurses, etc.),
   * Flyers and posters in health care facilities,
   * Distribution in the AddictLim network newsletter (pharmacists, nurses, social workers members),
   * Various: Liaison team, health delegate of the network, intranet site of the hospital, CCAS, AMPA, day care centers.
2. Conduct of a SCANVIR day in the non-conventional structure " Hors les murs " :

Each patient presenting during the screening day will have an individualized welcome.

Addictological and hepatological data will be collected throughout the process by the various workers on the individual Scanvir form (attached).

1. The patient accepts one or more of the examinations proposed as part of the routine care. After information, he/she does not object to the collection of his/her personal data.
2. One or more TRODs and a FibroScan® are performed by the nurse in charge of the care pathway and/or the facility.
3. Performing, by the biologist or the authorized person, the delocalized PCR in case of positive HCV TROD
4. Consultation with the hepatologist, who gives the results of the TROD and FibroScan® in a closed and dedicated place where the confidentiality of exchanges is guaranteed.
5. A written document with the results of the TROD and FibroScan® and GeneXpert is given to the patient.

Method for routine management of patients according to results :

1. HCV HBV HIV TROD are negative and FibroScan® > 7.1 KPa:

   The patient meets directly with the hepatologist to screen for risk factors for chronic liver disease (alcohol, medications ...).
2. The HCV HBV HIV TROD are negative and the FibroScan ® < 7.1 KPa :

   The nurse at the facility reviews with the patient the modes of transmission of the viruses and discusses with him/her risk reduction and harm reduction and what to do in case of recent exposure.
3. Positive HCV TROD:

   The hepatologist offers to do an immediate and on-site HCV RNA by delocalized PCR (GeneXpert). If the HCV RNA is positive, HCV treatment is started immediately (excluding comorbidity). An appointment is proposed 3 months after treatment to control the cure by delocalized PCR on site (RVS12)
4. HIV or HBV TROD positivity:

The hepatologist proposes to do immediately and on site a complete blood test (HIV serology, HBV serologies (HBsAg, HBcAb, HBsAb) by the nurse present, assesses other risk factors and schedules an appointment for the results and management.

For all situations, a prevention action to reduce the risks of transmission of HCV and HBV will be carried out at the same time.

An anti-viral B vaccination may be offered.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 and over
* Patient frequenting an unconventional structure "outside the walls" or referred by a professional in the care sector
* Patient who agreed to participate to the research

Exclusion Criteria:

* Patient doesn't agree to participate to the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People followed in unconventional structure care
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2022-12-09 (Estimated); Study Completion 2030-02-14 (Estimated)

PRIMARY OUTCOMES:
Number of RTDs performed compared to the number proposed | up to 10 years
  Evaluate the acceptability of simultaneous screening for viral hepatitis B, C and HIV among drug users in non-conventional structures using a dual method by RTDs and FibroScan®
Number of FibroScan® performed compared to the number proposed | up to 10 years
  Evaluate the acceptability of simultaneous screening for viral hepatitis B, C and HIV among drug users in non-conventional structures using a dual method by RTDs and FibroScan®

SECONDARY OUTCOMES:
Number of days actually completed and the number of participants per session | up to 10 years
  Evaluate the feasibility of simultaneous screening for viral hepatitis B, C and HIV in drug users in non-conventional structures using a dual screening method TROD and FibroScan®
Number and proportion of patients having accepted the immediate consultation with the hepatologist and/or with an addictologist | up to 10 years
  Evaluate the acceptability of risk reduction methods as part of the care pathway.
Number of patients who had social care | up to 10 years
  Evaluate the impact of screening in terms of patient care.
Number of anti-viral B vaccinations offered and carried out | up to 10 years
  Evaluate the impact of screening in terms of patient care.
Number of GeneXperts performed compared to the number proposed | up to 10 years
  Evaluate the impact of screening in terms of patient care.
The number and proportion of HCV or HBV antiviral treatments initiated in patients screened positive and having a therapeutic indication | up to 10 years
  Evaluate the impact of screening in terms of patient care.
Therapeutic compliance with anti-HCV treatments and sustained virological response rate in treated patients, | up to 10 years
  Evaluate the impact of screening in terms of patient care.
The absolute number and proportion of patients treated or not maintained in the care pathway in treated patients | up to 10 years
  Evaluate the impact of screening in terms of patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyne DEBETTE-GRATIEN, MD, Principal Investigator — Hôpital Dupuytren
Locations (1):
- Chu Limoges, Limoges, Haute Vienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Razavi H, Sanchez Gonzalez Y, Yuen C, Cornberg M. Global timing of hepatitis C virus elimination in high-income countries. Liver Int. 2020 Mar;40(3):522-529. doi: 10.1111/liv.14324. Epub 2019 Dec 23. PMID 31815353
- [Background] Tran A, Shili-Masmoudi S, Moga L, Chevaliez S, Luciani A, Ruiz I, Ganne-Carrie N, Bureau C, Bourliere M, de Ledinghen V. Non-invasive diagnosis and follow-up of chronic infection with Hepatitis C Virus. Clin Res Hepatol Gastroenterol. 2022 Jan;46(1):101771. doi: 10.1016/j.clinre.2021.101771. Epub 2021 Jul 28. PMID 34332129
- [Background] Pol S, Lagaye S. The remarkable history of the hepatitis C virus. Genes Immun. 2019 May;20(5):436-446. doi: 10.1038/s41435-019-0066-z. Epub 2019 Apr 25. PMID 31019253
- [Background] Brouard C, Pillonel J, Boussac M, de Ledinghen V, Rachas A, Silvain C, Lydie N, Chevaliez S, Pioche C, Durand J, Lot F, Delarocque-Astagneau E. French hepatitis C care cascade: substantial impact of direct-acting antivirals, but the road to elimination is still long. BMC Infect Dis. 2020 Oct 15;20(1):759. doi: 10.1186/s12879-020-05478-6. PMID 33059617
- [Background] Brouard C, Saboni L, Gautier A, Chevaliez S, Rahib D, Richard JB, Barin F, Larsen C, Sommen C, Pillonel J, Delarocque-Astagneau E, Lydie N, Lot F; 2016 Health Barometer Group. HCV and HBV prevalence based on home blood self-sampling and screening history in the general population in 2016: contribution to the new French screening strategy. BMC Infect Dis. 2019 Oct 28;19(1):896. doi: 10.1186/s12879-019-4493-2. PMID 31660879
- [Background] Bajis S, Grebely J, Hajarizadeh B, Applegate T, Marshall AD, Ellen Harrod M, Byrne J, Bath N, Read P, Edwards M, Gorton C, Hayllar J, Cock V, Peterson S, Thomson C, Weltman M, Jefferies M, Wood W, Haber P, Ezard N, Martinello M, Maher L, Dore GJ; LiveRLife Study Group. Hepatitis C virus testing, liver disease assessment and treatment uptake among people who inject drugs pre- and post-universal access to direct-acting antiviral treatment in Australia: The LiveRLife study. J Viral Hepat. 2020 Mar;27(3):281-293. doi: 10.1111/jvh.13233. Epub 2019 Dec 6. PMID 31698545
- [Background] Chevaliez S. Strategies for the improvement of HCV testing and diagnosis. Expert Rev Anti Infect Ther. 2019 May;17(5):341-347. doi: 10.1080/14787210.2019.1604221. Epub 2019 Apr 22. PMID 30950298
- [Background] Smookler D, Vanderhoff A, Biondi MJ, Valencia J, Ryan P, Karkada J, Hong R, Sattar I, Mandel E, Gjevori M, Casey J, Fletcher D, Shah H, Hansen BE, Capraru C, Janssen HLA, Lazarus JV, Feld JJ. Reducing Read Time of Point-of-Care Test Does Not Affect Detection of Hepatitis C Virus and Reduces Need for Reflex RNA. Clin Gastroenterol Hepatol. 2021 Jul;19(7):1451-1458.e4. doi: 10.1016/j.cgh.2020.07.058. Epub 2020 Aug 4. PMID 32763480
- [Derived] Debette-Gratien M, Francois S, Chevalier C, Alain S, Carrier P, Rigaud C, Abraham B, Burgevin AL, Courat L, Debenes B, Koffi J, Caux-Nussbaum E, Zattoni-Leroy J, Feuillet-Sow G, Dumont Q, Nubukpo P, Loustaud-Ratti V. Towards hepatitis C elimination in France: Scanvir, an effective model to test and treat drug users on dedicated days. J Viral Hepat. 2023 Apr;30(4):355-361. doi: 10.1111/jvh.13798. Epub 2023 Jan 11. PMID 36597183